CLINICAL TRIAL: NCT02136940
Title: A Phase 2a, Multicenter, Randomized, Double-masked, Placebo-controlled, Parallel-group Study of AMA0076 in Topical Ocular Formulation for Safety, Tolerability and Efficacy in Reduction of Intraocular Pressure in Subjects With Primary Open-angle Glaucoma or Ocular Hypertension
Brief Title: Multiple Dose-parallel-group Study of AMA0076 in Patients With Primary Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amakem, NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMA0076-S-202
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Glaucoma; Ocular Hypertension; Eye Disease
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AMA0076 0.1% (Experimental): Eligible subjects who meet the inclusion/exclusion criteria will be randomized to active or placebo (vehicle) in a 1:1:1:1 allocation ratio.
  Interventions: Drug: AMA0076
- AMA0076 0.25% (Experimental): Eligible subjects who meet the inclusion/exclusion criteria will be randomized to active or placebo (vehicle) in a 1:1:1:1 allocation ratio.
  Interventions: Drug: AMA0076
- AMA0076 0.50% (Experimental): Eligible subjects who meet the inclusion/exclusion criteria will be randomized to active or placebo (vehicle) in a 1:1:1:1 allocation ratio.
  Interventions: Drug: AMA0076
- Placebo (Placebo Comparator): Eligible subjects who meet the inclusion/exclusion criteria will be randomized to active or placebo (vehicle) in a 1:1:1:1 allocation ratio.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMA0076
  Arms: AMA0076 0.1%; AMA0076 0.25%; AMA0076 0.50%
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this parallel group study is to evaluate the safety, tolerability and efficacy of AMA0076 in reduction of intraocular pressure in subjects with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults 30-85 years of age.
* Diagnosis of either POAG or OHT in both eyes.
* Not receiving medication for IOP, or able to stop such medication for a washout period and the duration of the study without significant risk of adverse consequences related to glaucomatous disease.
* Elevated IOP (≥ 24 and ≤ 33 mm Hg at 8 AM and ≥ 21 and ≤ 33 mm Hg at 10 AM on Screening Two visit and Baseline visit in one or both eyes off treatment [after a washout phase in those subjects who were receiving ocular hypotensive therapy]).

Exclusion Criteria:

Ophthalmic exclusion criteria:

* Uncontrolled intraocular hypertension defined as > 33 mm Hg in either eye at either of the screening/baseline visits (after a washout phase in those subjects who were currently receiving ocular hypotensive therapy).
* Receiving more than one medication for IOP in either eye at time of screening.
* Abnormal central corneal thickness.
* BCVA worse than 20/200 (logMAR 1.0) in either eye
* Significant visual field loss.
* Acute angle-closure glaucoma or appositional or very narrow anterior chamber angle in either eye.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in mean diurnal intraocular pressure | 4 weeks

SECONDARY OUTCOMES:
Mean, mean change and percent change from baseline in intraocular pressure in both mean diurnal intraocular pressure and intraocular pressure at equivalent diurnal time points. | 4 weeks
Compare the safety and tolerability of topically administered AMA0076 compared to vehicle, by evaluation of safety variables | 4 weeks
  Evaluation of safety variables including eye exam findings (best corrected visual acuity, biomicroscopy [including grading of conjunctival hyperemia], dilated fundus examination) adverse events, discontinuations due to adverse events, serious adverse events, and vital signs.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Artesia Clinical - Site 11, Artesia, California
  - Inglewood Clinical Site - Site 15, Inglewood, California
  - Petaluma Clinical Site - Site 17, Petaluma, California
  - Morrow Clinical Site - Site13, Morrow, Georgia
  - Roswell Clinical Site - Site 18, Roswell, Georgia
  - Rochester Clinical Site - Site 12, Rochester, New York
  - Slingerlands Clinical Site - Site 19, Slingerlands, New York
  - Charlotte Clinical Site - Site 14, Charlotte, North Carolina
  - High Point Clinical Site - Site 16, High Point, North Carolina